CLINICAL TRIAL: NCT05088083
Title: Single-arm Study of Paclitaxel-Coated Percutaneous Transluminal Angioplasty (PTA) Balloon for the Treatment of Obstructive Lesions in the Native Arteriovenous Dialysis Fistulae (AVF)
Brief Title: Paclitaxel-Coated Balloon for the Treatment of AVF
Acronym: AVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Zylox Medical Device Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V1.0
Record Dates: First submitted 2021-09-20; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Arteriovenous Fistula
Keywords: DCB
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DCB Treatment Group (Experimental): Subjects treated with DCB
  Interventions: Device: Paclitaxel-Coated Percutaneous Transluminal Angioplasty (PTA) Balloon

INTERVENTIONS:
Device: Paclitaxel-Coated Percutaneous Transluminal Angioplasty (PTA) Balloon — After predilation, using drug-coated balloon catheter to cover the whole treated segment
  Other Names: Zylox

SUMMARY:
To evaluate the safety and efficacy of the Zylox Drug Coated Balloon (DCB) for treatment of subjects presenting with de novo or non-stented restenotic obstructive lesion of native arteriovenous dialysis fistulae (AVF) in the upper extremity in China.

ELIGIBILITY:
Inclusion Criteria:

* Age during 18-85 years old
* Arteriovenous fistula is matured and has undergone one or more hemodialysis sessions
* Venous stenosis of the AV fistula
* target lesion has stenosis ≥50% evidenced by angiography. and have at least one symptom of these：1,the venous pressure increased significantly during dialysis. 2,abnormal physical examination. 3,Decrease in blood flow
* the length of target lesion ≤100mm
* Patient able to give informed consent
* residual stenosis ≤30% after predilation

Exclusion Criteria:

* Women who are breastfeeding, pregnant or are intending to become pregnant
* AVF located at lower limbs
* Two or more than two stenosis at the target vessel.
* Obstruction of central venous return
* ISR
* AVF with acute thrombosis requiring lysis or thrombectomy in 30 days
* Vascular access has surgery in 30 days or intending to undergo a surgery
* Known hypersensitivity to aspirin, heparin, clopidogrel,paclitaxel, contrast medium, etc.
* Patients undergoing immunotherapy or suspected / confirmed vasculitis
* Patients with history of blood coagulation dysfunction and history of thrombocytopenic purpura
* Vascular access infection or systemic active infection
* Patients's life expectancy is less than 12 months
* Renal transplantation has been planned or converted to peritoneal dialysis
* Other medical conditions that lead to researchers who believe that patients may not be able to follow the trial program
* Involved in other drugs, biology, medical device research, or has been involved in other similar products clinical Test

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
primary patency of target lesion in 6 months | 6 months
  Primary Patency is defined as the freedom of reintervention for the target lesion,including: 1)clinical driven target lesion reintervention; 2) PSVR< 2.4

SECONDARY OUTCOMES:
Device Success | Time of procedure
  Successful delivery to the target lesion, deployment, and retrieval at index procedure
Clinical Success | From the time of the index procedure to the first successful dialysis session after index procedure. Typically, this is within 1 week of index procedure.
  The resumption of dialysis for at least one session after the index procedure
Procedural Success | 2 weeks
  Maintenance of patency (≤30% residual stenosis) in the absence of peri-procedural serious adverse device effect (SADE).

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhang, Principal Investigator — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No